CLINICAL TRIAL: NCT04097366
Title: Breast Screening - Risk Adaptive Imaging for Density
Acronym: BRAID
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cancer Research UK (Other); GE Healthcare (Industry); Queen Mary University of London (Other); Public Health England (Other Government)
Responsible Party: Principal Investigator, Fiona J Gilbert, Professor of Radiology and Head of Department, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A095053
Record Dates: First submitted 2019-09-09; First posted 2019-09-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of Care (No Intervention): Control arm, no supplementary imaging is given. Participants have mammographic screening 3-yearly as per current standard of are.
- Abbreviated MRI (ABB-MRI) (Active Comparator): Supplementary imaging with abbreviated MRI at study entry and 18 months after baseline mammogram.
  Interventions: Diagnostic Test: ABB-MRI
- Automated Breast Ultrasound (ABUS) (Active Comparator): Supplementary imaging with automated breast ultrasound at study entry and 18 months after baseline mammogram.
  Interventions: Diagnostic Test: ABUS
- Contrast Enhanced Mammography (CEM) (Active Comparator): Supplementary imaging with contrast enhanced spectral mammography at study entry and 18 months after baseline mammogram.
  Interventions: Diagnostic Test: CEM

INTERVENTIONS:
Diagnostic Test: ABUS — Automated whole breast ultrasound (ABUS) is undertaken with a large transducer panel placed on the breast in three positions. Resultant images are combined to make a 3D image of the breast.
  Other Names: Whole Breast Ultrasound; Automated Breast Ultrasound
  Arms: Automated Breast Ultrasound (ABUS)
Diagnostic Test: CEM — A high kV and a low kV image is taken in two standard views of each breast following the intravenous injection of an iodinated contrast agent.
  Other Names: Contrast Enhanced Mammography
  Arms: Contrast Enhanced Mammography (CEM)
Diagnostic Test: ABB-MRI — ABB-MRI is a shorter version of breast MRI. Standard T1W pre and post contrast images are acquired. A MIP and post-contrast T1 weighted image are read.
  Other Names: Abbreviated Magnetic Resonance Imaging; Abridged MRI; Abbreviated Protocol MRI; Abbreviated Breast MRII
  Arms: Abbreviated MRI (ABB-MRI)

SUMMARY:
BRAID is a randomised, multi-centre study assessing the impact of supplementary imaging in the detection of breast cancer in women participating in the UK national breast screening programme who have dense breast tissue.

DETAILED DESCRIPTION:
Breast density is a measure of the amount of fibroglandular tissue and is a risk factor for breast cancer. Women with extremely dense breasts are at 4-fold increased breast cancer risk compared to women with 'fatty' breasts. High breast density reduces the sensitivity of mammography increasing the probability of the test missing a cancer. Women with dense breasts have their cancers found when the cancer is larger as they present with interval cancers or their cancers are not detected until the next screening round at a later stage.

The UK national breast screening programme (NHS BSP) offers all women aged 50-70 screening with 3-yearly mammograms. It aims to reduce breast cancer mortality by 20% by detecting small cancers thereby reducing the number of late stage diagnoses. However only 53% of the cancers being detected are small (<15mm). This is partly due to masking of cancers by dense breast tissue.

This trial addresses how best to screen women with dense breasts for breast cancer. BRAID will randomise women whose recent screening normal mammogram shows that they have dense breasts to either standard of care (no supplementary imaging) or supplementary imaging with abbreviated MRI (ABB-MRI), automated whole breast ultrasound (ABUS) or contrast enhanced spectral mammography (CEM). These imaging techniques have been shown to be more sensitive than mammography at detecting cancers in dense breast tissue. Our hypothesis is that more cancers will be detected at an earlier stage with supplemental imaging.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Willing and able to comply with the scheduled study visits, tests and other procedures
* Female
* Screening mammogram that is either normal or being recalled for assessment
* Increased breast density identified on current screening mammogram examination (BIRADS C or D)

  * If BIRADS C the reporting radiologist should use clinical judgement as to eligibility, there should be a high chance of a cancer being masked in this participant
  * All BIRADS D will be eligible
* Aged 50-70 and eligible for 3-yearly NHS breast screening

Exclusion Criteria:

* Known BRCA carrier or ≥50% risk of being a carrier
* Unable to give informed consent
* Breast implant(s)
* Unable to be followed-up for the study duration
* Current participation in another interventional breast screening trial (Including but not limited to MyPeBS)
* Participated in part A of the BRAID study
* Pregnant or breast feeding

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9000 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cancer detection rate in each arm | 42 months after mammogram at study entry
  All cancers (detected or interval) in each arm over a three year period will be collected.

SECONDARY OUTCOMES:
Incidence of stage II or worse cancers over the period of observation | 42 months after last participant entered
  size, lymph node status, metastatic status
The sensitivity and specificity of supplemental imaging with ABB-MRI, CESM and ABUS with standard 2D FFDM. | 6 months after mammogram at study entry
  Analysis will include: Detection rate of all breast cancers, Detection rate of all breast cancers by stage; Detection rate of all breast cancers by biological type; Detection rate of all breast cancers by size; Recall rates at prevalent round
The sensitivity and specificity of supplemental imaging with ABB-MRI, CESM and ABUS with standard 2D FFDM. | 21 months after mammogram at study entry
  Analysis will include: Detection rate of all breast cancers, Detection rate of all breast cancers by stage; Detection rate of all breast cancers by biological type; Detection rate of all breast cancers by size; Recall rates
The sensitivity and specificity of supplemental imaging with ABB-MRI, CESM and ABUS with standard 2D FFDM. | 42 months after last participant entered
  Analysis will include: Detection rate of all breast cancers, Detection rate of all breast cancers by stage; Detection rate of all breast cancers by biological type; Detection rate of all breast cancers by size; Recall rates at incident round; Interval cancer rate; Stage of interval cancers; Size of interval cancers
Reading time of each examination | 1 year
  Average time and range for each modality. (Seconds).
Automated breast density measurements compared with reader assessment | Baseline
  Percentage density.
The risk of developing breast cancer as assessed by the BOADICEA model | 72 months After last participant entered
  Percentage 5 year risk, percentage lifetime risk.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Gilbert, Principal Investigator — University of Cambridge
Locations (10):
- United Kingdom (10):
  - Tayside Health Board, Ninewells Hospital, Dundee, Dundee
  - Greater Glasgow Health Board, Gartnavel Royal Hospital, Glasgow, Glasgow
  - University Hospitals of Leicester, Leicester Royal Infirmary, Leicester, Leicestershire
  - Barts Health NHS Trust, Royal London Hospital, London, London
  - Royal Free London NHS Foundation Trust, London, London
  - Nottingham University Hospitals NHS Trust, City Hospital, Nottingham, Nottinghamshire
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - The Leeds Teaching Hospitals NHS Trust, Leeds
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilbert FJ, Payne NR, Allajbeu I, Yit L, Vinnicombe S, Lyburn I, Sharma N, Teh W, James J, Seth A, Suaris T, Aggarwal R, Al-Attar M, Savaridas S, Antoniou A, Pharoah P, Duffy S. Comparison of supplemental breast cancer imaging techniques-interim results from the BRAID randomised controlled trial. Lancet. 2025 May 31;405(10493):1935-1944. doi: 10.1016/S0140-6736(25)00582-3. Epub 2025 May 21. PMID 40412427